CLINICAL TRIAL: NCT04586959
Title: Uterine Manipulation During Minimally Invasive Surgery for Early Stage Endometrial Cancer
Acronym: MAN-U
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anthony Costales, MD (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Anthony Costales, MD, Assistant Professor Obstetrics & Gynecology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-46373
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: ENDOMETRIAL CANCER
Keywords: endometrial; cancer; uterine; manipulator
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: A prospective multi-center non-inferiority randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surgery With UM (Arm MAN UA) (Experimental): Subjects that undergo a MIS approach with a uterine manipulator (experimental arm)
  Interventions: Device: Surgery with UM
- Surgery Without UM (Arm Control) (Active Comparator): Subjects that undergo a MIS approach without a uterine manipulator (control arm)
  Interventions: Device: Surgery without UM

INTERVENTIONS:
Device: Surgery with UM — The experimental group will have MIS with the placement of a uterine manipulator
  Arms: Surgery With UM (Arm MAN UA)
Device: Surgery without UM — The control group will have MIS without the placement of a uterine manipulator
  Arms: Surgery Without UM (Arm Control)

SUMMARY:
This is a prospective, multi-center, randomized non-inferiority phase III study to evaluate if patients undergoing a minimally invasive surgery for early stage uterine cancer have cancer cells in the fluid that is obtained at the time of their surgery when a uterine manipulator is placed versus patients who do not have a uterine manipulator placed.

DETAILED DESCRIPTION:
In most cases, patients who have early stage endometrial cancer undergo a surgery to remove the uterus, cervix, tubes, ovaries, and occasionally lymph nodes. This is usually done through a minimally invasive (not a large incision) surgery. To accomplish this, the uterus needs to be manipulated (moved around) to help the surgeon complete your surgery. This is usually done with a device called a uterine manipulator and the majority of surgeons use this device in any patient undergoing a minimally invasive hysterectomy (removal of the uterus and cervix).

Even though the majority of surgeons use a manipulator, there are some surgeons who believe there is a possibility that cancer cells inside the uterus can be spilled into the abdomen through the fallopian tubes. This may cause a higher risk of spreading the cancer and or of the cancer coming back.

Currently, there are very limited research studies directly looking at whether the uterine manipulator may cause these cells to appear in the abdomen.

The purpose of this study is to see if patients undergoing a minimally invasive surgery for early stage uterine cancer have cancer cells in the fluid that is obtained at the time of their surgery when a uterine manipulator is placed versus patients who do not have a uterine manipulator placed.

A computer program will randomly assign the subjects to one of two groups. One group will have minimally invasive surgery with the use of a uterine manipulator and the other group will have minimally invasive surgery without the use of a uterine manipulator.

Researchers will use the information from this study to decide how best to take care of patients undergoing minimally invasive surgery for uterine cancer.

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered eligible for inclusion in this study if all the following criteria are met:

1. Patient must be greater than or equal to 18 years old.
2. Suspected clinically early stage endometrial cancer of any histology (endometrioid, mixed, serous, clear-cell, carcinosarcomas, mucinous)
3. Pre-operative imaging not suggestive of extra-uterine disease, if obtained pre-operatively.
4. CA 125 testing is optional but, if obtained, must be within lab normal values. 5. ECOG performance status 0-2 (see appendix 1).

6. Signed informed consent and ability to comply with follow-up. 7. Per the opinion of the treating investigator, the patient must be a suitable candidate for the MIS surgical procedure.

Exclusion Criteria:

A subject must not have any of the following criteria:

1. Planned laparotomic hysterectomy
2. On progesterone therapy to treat their endometrial cancer
3. Any prior pelvic irradiation

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 278 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Positive peritoneal cytology (PC) | Immediately after uterine manipulator placement in the manipulator group or prior to the initiation of the hysterectomy procedure in the non-manipulator group
  Positive PC is defined as the presence of malignant cells in the peritoneal cytology specimen.

SECONDARY OUTCOMES:
Post-operative positive PC | Immediately after closure of the vaginal cuff
  Positive PC is defined as the presence of malignant cells in the peritoneal cytology specimen.
Lymphovascular space invasion (LVSI) | During surgery
  LVSI is defined as the presence of tumor cells within a definite endothelial-lined space (lymphatics or blood vessels) at the advancing edge of the tumor as it invades the myometrium, within an endometrial polyp, or within the endometrial stroma.
Percentage of myometrial invasion (MI) | During surgery
  Defined as the % of invasion into the myometrium from the endomyometrial junction
Extent of lymph node metastases | During surgery
  Defined as presence of isolated tumor cells (ITC - <0.2 mm), or micrometastasis (mm - 0.2 - 2 mm), or macrometastasis (MM - > 2 mm), whichever is greater.
Operative time | 1 day
  Defined as time from start of operation to closure of skin in minutes as documented in the electronic medical record
Surgical morbidity | Intra-operative and up to 30 days post-surgery
  Surgical morbidity (CTCAE v5.0) grade 3 and higher, or any grade of the following adverse events: colonic fistula, colonic perforation, enterovesical fistula, gastrointestinal fistula, ileus, intra-abdominal hemorrhage, rectal fistula, rectal perforation, small intestinal perforation, abdominal infection, pelvic infection, vaginal infection, intra-operative arterial injury, venous injury, intra-operative gastrointestinal injury, intra-operative hemorrhage, intra-operative neurological injury, intra-operative urinary injury, and post-operative hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Costales, MD, Principal Investigator — Baylor College of Medicine
Locations (5):
- United States (5):
  - Cleveland Clinic, Cleveland, Ohio
  - Baylor College of Medicine- McNair Campus, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No